CLINICAL TRIAL: NCT00389831
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Proof-of-concept Trial to Assess the Efficacy, Safety and Tolerability of Ascending Doses of Rotigotine Nasal Spray for the Acute Treatment of RLS Symptoms in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: Efficacy, Safety and Tolerability of Rotigotine Nasal Spray for the Acute Treatment of RLS Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0879; 2006-001937-17 (EudraCT Number)
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2011-02

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Rotigotine nasal spray; Efficacy, safety and tolerability; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects receiving a single dose of placebo nasal spray on all 4 treatment days
  Interventions: Other: Placebo Nasal Spray
- Rotigotine Nasal Spray (Experimental): Subjects receiving doses of placebo nasal spray on Day 1 or Day 2, Rotigotine nasal spray 62µg on Day 1 or Day 2, Rotigotine nasal spray 124µg on Day 3, and Rotigotine nasal spray 247µg on Day 4
  Interventions: Drug: Rotigotine Nasal Spray

INTERVENTIONS:
Drug: Rotigotine Nasal Spray — Daily single dose of 62µg, 124µg, and 247µg rotigotine delivered as single puff of nasal spray solution
  Other Names: SPM937
  Arms: Rotigotine Nasal Spray
Other: Placebo Nasal Spray — Daily single dose of placebo delivered as single puff of nasal spray solution
  Arms: Placebo

SUMMARY:
The main objective of this phase 2a proof-of-concept trial is to assess the efficacy of rotigotine nasal spray in ascending doses in subjects with idiopathic Restless Legs Syndrome.

DETAILED DESCRIPTION:
Each patient of the placebo and rotigotine group performed an Eligibility Assessment, as well 4 treatment days at which subjects performed a repeated 'Suggested Immobilization Test' (SIT) during a 30min pre-dose and a 4 hours post-dose period. During these periods the severity of RLS symptoms in the legs was assessed by the subject using a numeric symptom severity scale.

In addition the leg movements were measured by actigraphy to assess the Periodic Leg Movement Index during Wakefulness (PLMWI, PLM per hour). Subjects applied a single dose of treatment on each treatment day (placebo nasal spray or rotigotine nasal spray in 3 ascending doses).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with idiopathic RLS, who are responding to an ongoing L-dopa treatment

Exclusion Criteria:

* Patients with secondary RLS or clinically relevant concomitant diseases or medical conditions are excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Raetz, Study Director — Schwarz BioSciences GmbH
Locations (1):
- Schwarz BioSciences GmbH, Monheim, Germany

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rotigotine Nasal Spray
Started | 10 | 34
Completed | 10 | 27
Not Completed | 0 | 7
Not completed — Lack of Efficacy | 0 | 2
Not completed — Did not receive treatment. | 0 | 2
Not completed — Other reasons | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine Nasal Spray | Total
Number analyzed (Participants) | 10 | 34 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 33 | 42
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (5.40) | 52.9 (7.78) | 53.5 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 21 | 29
  Male | 2 | 13 | 15
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 34 | 44

OUTCOME MEASURES:

1. Primary Outcome: Average Numeric Symptom Severity Score After Single Dose of Rotigotine Nasal Spray or Matching Placebo
Description: Subjects rate the severity of the RLS symptoms at the start of each pre dose and post dose Suggested Immobilization Test (SIT-0 to SIT-6) and every 5min during each SIT, using a numeric symptoms severity scale, where 0=not severe and 10=very severe.
Time Frame: 4 hours post-treatment period at each treatment day
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo - Day 1: Subjects randomized to placebo treatment arm receiving a single dose of placebo nasal spray on Day 1.
- Placebo - Day 2: Subjects randomized to placebo treatment arm receiving a single dose of placebo nasal spray on Day 2.
- Placebo - Day 3: Subjects randomized to placebo treatment arm receiving a single dose of placebo nasal spray on Day 3.
- Placebo - Day 4: Subjects randomized to placebo treatment arm receiving a single dose of placebo nasal spray on Day 4.
- Rotigotine Nasal Spray - Placebo: Subjects randomized to rotigotine nasal spray arm receiving a single dose of placebo nasal spray on Day 1 or Day 2.
- Rotigotine Nasal Spray - Rotigotine 62µg: Subjects randomized to rotigotine nasal spray arm receiving a single dose of rotigotine 62µg nasal spray on Day 1 or Day 2.
- Rotigotine Nasal Spray - Rotigotine 124µg: Subjects randomized to rotigotine nasal spray arm receiving a single dose of rotigotine 124µg nasal spray on Day 3.
- Rotigotine Nasal Spray - Rotigotine 247µg: Subjects randomized to rotigotine nasal spray arm receiving a single dose of rotigotine 247µg nasal spray on Day 4.
Arm/Group | Placebo - Day 1 | Placebo - Day 2 | Placebo - Day 3 | Placebo - Day 4 | Rotigotine Nasal Spray - Placebo | Rotigotine Nasal Spray - Rotigotine 62µg | Rotigotine Nasal Spray - Rotigotine 124µg | Rotigotine Nasal Spray - Rotigotine 247µg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 31 | 31 | 28 | 28
score on a scale | 2.6 (1.76) | 2.2 (1.44) | 2.5 (2.03) | 2.0 (1.65) | 2.9 (1.99) | 2.7 (1.84) | 2.0 (1.14) | 1.5 (1.21)

2. Primary Outcome: Average PLMWI (Periodic Leg Movement Index During Wakefulness) After Single Dose of Rotigotine Nasal Spray or Matching Placebo.
Description: The Periodic Limb Movement (PLM) during Wakefulness Index (PLMWI) measures the number of limb movements per hour and indicates the frequency of PLMs when the subject is awake and the degree of motor symptoms of the disorder during wake time. No movements would result in a score of 0 PLM per hour. Outcome is the average movements per hour in the 4 hour post-dose period per subject.
Time Frame: 4 hours post-treatment period at each treatment day
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: PLM per hour
Arm/Group | Placebo - Day 1 | Placebo - Day 2 | Placebo - Day 3 | Placebo - Day 4 | Rotigotine Nasal Spray - Placebo | Rotigotine Nasal Spray - Rotigotine 62µg | Rotigotine Nasal Spray - Rotigotine 124µg | Rotigotine Nasal Spray - Rotigotine 247µg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 31 | 31 | 27 | 28
PLM per hour | 37.8 (35.10) | 22.6 (28.36) | 34.9 (39.78) | 19.0 (23.60) | 28.7 (29.91) | 25.4 (25.14) | 26.2 (22.78) | 20.2 (21.70)

ADVERSE EVENTS:
Groups:
- Placebo - Day 1: Subjects randomized to placebo treatment group, receiving a single dose of placebo nasal spray on Day 1.
- Placebo - Day 2: Subjects randomized to placebo treatment group, receiving a single dose of placebo nasal spray on Day 2.
- Placebo - Day 3: Subjects randomized to placebo treatment group, receiving a single dose of placebo nasal spray on Day 3.
- Placebo - Day 4: Subjects randomized to placebo treatment group, receiving a single dose of placebo nasal spray on Day 4.
Arm/Group | Placebo - Day 1 | Placebo - Day 2 | Placebo - Day 3 | Placebo - Day 4 | Rotigotine Nasal Spray - Placebo | Rotigotine Nasal Spray - Rotigotine 62µg | Rotigotine Nasal Spray - Rotigotine 124µg | Rotigotine Nasal Spray - Rotigotine 247µg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/31 | 0/31 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10 | 2/10 | 2/10 | 16/31 | 14/31 | 10/28 | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Day 1 (N=10) | Placebo - Day 2 (N=10) | Placebo - Day 3 (N=10) | Placebo - Day 4 (N=10) | Rotigotine Nasal Spray - Placebo (N=31) | Rotigotine Nasal Spray - Rotigotine 62µg (N=31) | Rotigotine Nasal Spray - Rotigotine 124µg (N=28) | Rotigotine Nasal Spray - Rotigotine 247µg (N=28)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteria urine identified (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 9 (10) | 5 (6) | 3 (4) | 3 (3)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.